CLINICAL TRIAL: NCT02140125
Title: Phase I Study of ASP2408 -Subcutaneous Single-dose, Placebo-controlled Study in Non-elderly Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Safety of ASP2408 After Subcutaneous Administration to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2408-CL-9101
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Healthy; Pharmacokinetics of ASP2408
Keywords: ASP2408
MeSH Terms: interventions — ASP2408

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP2408 low dose group (Experimental)
  Interventions: Drug: ASP2408
- ASP2408 middle dose group (Experimental)
  Interventions: Drug: ASP2408
- ASP2408 high dose group (Experimental)
  Interventions: Drug: ASP2408
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2408 — subcutaneous administration
  Arms: ASP2408 high dose group; ASP2408 low dose group; ASP2408 middle dose group
Drug: Placebo — subcutaneous administration
  Arms: Placebo group

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of single subcutaneous dose of ASP2408 in non-elderly healthy adult male subjects. The pharmacodynamics of ASP2408 is also being evaluated.

DETAILED DESCRIPTION:
This clinical study will be conducted as a double-blind, placebo-controlled, single ascending subcutaneous dose study. As shown in the table below, the study will be conducted using 3 cohorts, to which a total of 24 subjects will be randomly assigned (18 subjects receiving ASP2408 and 6 subjects receiving placebo). Each cohort will consist of 8 subjects, who will be randomly assigned to either the ASP2408 group or the placebo group at the ratio of 3 to 1.

Each subject will need to be hospitalized until Day 8 (start date of study drug administration will be regarded as Day 1) and will be observed until Day 90. The investigator or subinvestigator will carefully observe each subject for any sign or symptom of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* BMI (at screening): ≥ 17.6 kg/m2, < 26.4 kg/m2
* Healthy, as judged by the investigator or subinvestigator based on the results of medical examination (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospitalization (Day -2) to immediately before study drug administration
* Subjects who agree to use effective contraception until 90 days after study drug administration

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before the study or is scheduled to receive any investigational drugs
* Donated 400 mL of whole blood within 90 days before the study or during the period from the screening, 200 mL of whole blood within 30 days, or blood components within 14 days before the study, or is scheduled to donate 400 mL of whole blood or blood components
* Received medication within 7 days before hospitalization (Day -2) or is scheduled to receive medication
* Received systemic medications influencing immune functions (e.g., steroids, tacrolimus hydrate, anticancer drugs, and biological products) within 365 days before study drug administration
* Received a live virus vaccine (e.g., BCG, polio, measles, and rubella) within 180 days before study drug administration, or cannot agree not to receive these vaccines for 180 days after study drug administration
* Received a live virus vaccine (e.g., BCG, polio, measles, and rubella) within 180 days before study drug administration, or cannot agree not to receive these vaccines for 180 days after study drug administration
* A deviation from the normal range of blood pressure, pulse rate, body temperature, or standard 12-lead ECG (see Table 3.3-1) at screening or the day before study drug administration (Day -1)
* Any deviation of the normal ranges in laboratory tests before study drug administration
* Failure to meet any criteria for standard 12-lead ECG for QT assessment at screening
* A positive result for tuberculosis test
* Concurrent or history of drug allergies, anaphylaxis, or severe allergic reaction
* Upper GI disease
* Concurrent or previous hepatic disease (e.g., viral hepatitis and drug-induced liver injury)
* Concurrent or previous heart disease (e.g., congestive heart failure, angina pectoris, and arrhythmia requiring treatment)
* Concurrent or previous respiratory disease (e.g., bronchial asthma and chronic bronchitis; except for a history of childhood asthma)
* Previous operation of gut excision
* Concurrent or previous renal disease (e.g., acute renal failure, glomerulonephritis, and interstitial nephritis; except for a history of calculus)
* Concurrent or previous endocrine disease (e.g., hyperthyroid, abnormality of growth hormone)
* Concurrent or previous cerebrovascular disorder (e.g., cerebral infarction)
* Concurrent or previous malignant tumor
* Concurrent or previous serious infection (e.g., sepsis, pneumonia requiring hospitalization, and pyelonephritis)

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, lab tests, and 12-lead ECG | Up to 90 days after administration

SECONDARY OUTCOMES:
Pharmacokinetics of serum ASP2408 | On day-1, day-2, day-3, day-4, day-5, day-6, day-7, day-8, day-9, day-11, day-13, day-15, day-22, day-29 day-43, day-60 and day-90
  The pharmacokinetic analysis employed non-compartmental methods using serum concentrations of ASP2408. The following pharmacokinetic parameters were estimated: AUCinf, AUClast, Cmax, CL/F, tmax, t1/2, and Vz/F.
CD80/CD86 receptor occupancy | On day-1, day-2, day-3, day-5, day-8, day 15, day-22, day-29 and day-90
Total lymphocyte count | On day-1, day-2, day-3, day-5, day-8, day 15, day-22, day-29 and day-90
Peripheral blood lymphocyte subset | On day-1, day-2, day-3, day-5, day-8, day 15, day-22, day-29 and day-90

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan